CLINICAL TRIAL: NCT05230212
Title: Cognitive Function in Response to a Pecan-Enriched Meal
Brief Title: Pecan Consumption and Cognitive Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Jamie Cooper, PhD, Professor, University of Georgia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: PROJECT00004889
Record Dates: First submitted 2022-01-22; First posted 2022-02-08 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: This trial will be a double-blinded, randomized, cross-over design. There will be 2 testing visits in which each participant will be randomized to receive either the control (cream) shake or the pecan shake at visit 1; they will receive the opposing shake at visit 2. There will be a 6-8 day washout period between visit 1 and visit 2.
Who Masked: Participant, Investigator
Masking Description: Involved researchers and participants are blinded to which breakfast shake they are administering and/or receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pecan Breakfast Shake (Experimental): Participants will be given a breakfast shake consisting primarily of pecans, and 1% milk.
  Interventions: Other: Pecan Breakfast Shake
- Cream Breakfast Shake (Active Comparator): Participants will be given a breakfast shake consisting primarily of heavy whipping cream.
  Interventions: Other: Cream Breakfast Shake

INTERVENTIONS:
Other: Pecan Breakfast Shake — The pecan breakfast shake contains 68 grams of blended raw pecans. Participants will consume this shake at either visit 1 or visit 2 depending on randomization procedures.
  Arms: Pecan Breakfast Shake
Other: Cream Breakfast Shake — The cream breakfast shake contains 138 grams of heavy whipping cream. Participants will consume this shake at either visit 1 or visit 2 depending on randomization procedures.
  Arms: Cream Breakfast Shake

SUMMARY:
Human cognitive function is affected by age-related changes, with some areas beginning to decline in mid-adulthood and worsening with age. However, there is evidence that dietary interventions or the incorporation of certain healthy foods or nutrients, into the diet can have protective effects against cognitive decline. These foods include nutrients such as polyunsaturated fats, vitamins E and C, and polyphenols. Pecans are a rich source of polyunsaturated fatty acids, antioxidants (including polyphenols), and vitamin E. Pecans contain more total phenols than any other tree nut suggesting that they may be an ideal bioactive food to enhance cognitive performance; however, the relationship between pecan consumption and cognitive functioning has never been assessed. The overall goal behind this research is to determine the relationship between antioxidant-rich pecans and cognitive functioning in a postprandial state.

DETAILED DESCRIPTION:
This trial will be a double-blinded, randomized, cross-over design in humans. There will be two study visits for two different test meals administered in random order. The two testing visits (v1 and v2) include blood draws and repetitions of the cognitive battery after consuming one of the two different test meals containing 1% milk, Nesquik, and either: 1) pecans, or 2) heavy whipping cream. There will be a 6-8 day washout period between each study visit.

Hypothesis: Investigators hypothesize that the pecan-enriched meal will 1.) improve performance on select measures of postprandial cognitive functioning (such as executive functioning, memory, learning, attention, and processing speed) 2.) improve postprandial markers of glycemic control, inflammation, antioxidant capacity, coagulation potential, and 3.) present a similar suppression of subjective appetite compared to the isocaloric, control meal that does not contain pecans.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 30-years-old
* Healthy individuals
* Men and Women
* Normal body mass index (BMI) (18.5-24.9kg/m2). If BMI is 25 or greater, subjects can still qualify if their body fat percentage falls within healthy ranges defined as Men: 5-20%, and Women: 15-30% [22]
* Individuals with normal or corrected to normal vision
* Low-risk alcohol use as assessed by the AUDIT questionnaire (need a score of 7 or lower)
* No or minimal depression symptoms as indicated by the Beck's Depression Inventory (need a score of 9 or lower)
* Cognitive competence for education level and age as measured by the Mini-Mental State Examination (need a score of 26 or higher)

Exclusion Criteria:

* All chronic diseases (including, but not limited to, renal or bowel diseases, cardiovascular disease, and any form of diabetes)
* Known neurological, cognitive, or psychiatric conditions (including, but not limited to, mood disorders, anxiety disorders, and depression)
* Prescription medication use (with the exception of female contraception methods)
* Dietary supplement use (including, but not limited to, multivitamins and fish oil supplements)
* Alcohol intake >3 drinks/d for males or >2 drinks/d for females
* Diagnosis of ADHD or a learning difficulty (including, but not limited to, dyslexia)
* History of head injury (defined as loss of consciousness more than 10 minutes)
* History of inflammatory disorders (including, but not limited to, migraines, stroke, hypertension, hypercoagulation, vascular disease, thyroid conditions, blood disorders, coagulation disorders)
* Food allergies/sensitivities to foods provided in this protocol including tree nuts, gluten, and or lactose/dairy
* Regular consumption of nuts and/or nut butters defined as consumption of >2 servings (60g) of tree nuts or nut butters (e.g., peanut butter, almond butter) per week
* High caffeine consumption, defined as >400mg/d
* Individuals adhering to special diets (including, but not limited to, the ketogenic diet, intermittent fasting, Atkins diet, vegan diet, vegetarian diet, or carbohydrate-restricted diets)
* Illicit drug use
* Smoking or use of tobacco products
* Color-blindness
* History of current renal or bowel disease
* Females who are currently pregnant or lactating
* Active individuals (defined as performing >5 hours/week of scheduled exercise)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2023-02-25 (Actual)

PRIMARY OUTCOMES:
Change in Alphabetic Working Memory, Choice Reaction Time, Digit Vigilance, N-back test, Word Recognition, Rapid Visual Information Processing, Picture Recognition, Immediate Word Recall, and Delayed Word Recall | Change from baseline to 4 hours postprandially
  Measured by Computerized Mental Performance Assessment System (COMPASS) computed scores of percent accuracy (total overall target stimuli/novel stimuli)
  Brain, Performance, and Nutrition Research Centre, Northumbria University
Change in Serial Subtractions, Immediate Word Recall, and Delayed Word Recall. | Change from baseline to 4 hours postprandially
  Measured by Computerized Mental Performance Assessment System (COMPASS) computed scores of the number of responses (total correct responses/error responses)
  Brain, Performance, and Nutrition Research Centre, Northumbria University
Change in Alphabetic Working Memory, Choice Reaction Time, Digit Vigilance, N-back, Picture Recognition, Rapid Visual Information Processing, Word Recognition. | Change from baseline to 4 hours postprandially
  Measured by Computerized Mental Performance Assessment System (COMPASS) computed scores of reaction time (msec) (overall, correct response, target stimuli, novel stimuli, number of false alarms, and number of missed sequences)
  Brain, Performance, and Nutrition Research Centre, Northumbria University

SECONDARY OUTCOMES:
Change in glucose and triglycerides | Change from baseline to 4 hours postprandially
  Blood samples will be collected to measure Glucose (mg/dL), Triglycerides (mg/dL)
Change in physiologic measures of appetite | Change from baseline to 4 hours postprandially
  Blood samples will be collected to measure Peptide YY (PYY) (pg/mL), Cholecystokinin (CCK) (pg/mL), Ghrelin (pg/mL), Glucagon-like Peptide 1 (GLP-1) (pg/mL), Gastric Inhibitory Peptide (GIP) (pg/mL), pancreatic peptide (PP) (pg/mL).
Change in lipid peroxidation | Change from baseline to 4 hours postprandially
  Malondialdehyde (MDA) (uM) measured via Thiobarbituric acid reactive substances (TBARS) assay.
Change in insulin | Change from baseline to 4 hours postprandially
  Insulin (uU/mL)
Change in non-esterified free fatty acids (NEFA) | Change from baseline to 4 hours postprandially
  NEFA (mEq/L)
Change in angiopoietin-like proteins-3 (ANGPTL3), angiopoietin-like-4 (ANGPTL4), and angiopoietin-like-8 (ANGPTL8) | Change from baseline to 4 hours postprandially
  ANGPTL-3 (pg/mL), ANGPTL-4 (pg/mL), ANGPTL-8 (pg/mL)
Change in subjective measures of appetite | Change from baseline to 4 hours postprandially. Also measured every hour for 10 hours after subject leaves the lab.
  Appetite Visual Analog Scale (VAS) (mm). The range of scores on the continuous VAS is 0-100 mm. Zero represents no hunger, fullness, prospective consumption, and desire to eat, while 100 represents the greatest feeling of these outcomes.
Change in total antioxidant capacity | Change from baseline to 4 hours postprandially
  Total antioxidant capacity (uM trolox equivalents) measured via Oxygen Radical Absorbance Capacity (ORAC) assay.
Change in oxidized low density lipoprotein (LDL) | Change from baseline to 4 hours postprandially
  Oxidized Low-Density Lipoprotein (ox-LDL) (mg/dL)

OTHER OUTCOMES:
Change in subjective measures of motivation | Change from baseline to 4 hours postprandially
  Motivation Visual Analog Scale (VAS) (mm). The range of scores on the continuous VAS is 0-100 mm. Zero represents no motivation while 100 represents the greatest feeling of this outcome.
Change in subjective measures of alertness, stress, and tranquility | Change from baseline to 4 hours postprandially
  Computerized Mental Performance Assessment System (COMPASS) - Brain, Performance, and Nutrition Research Centre, Northumbria University.
  Visual Analogue Mood Scales (VAMS) (mm). The range of scores on the continuous VAS is 0-100 mm. Zero represents lesser feeling of alertness, stress, and tranquility, while 100 represents the greatest feeling of these outcomes.
Change in subjective degree of sleepiness | Change from baseline to 4 hours postprandially
  Stanford Sleepiness Scale, in which the scale is rated from 1 to 7. A rating of 1 indicates feelings of being wide awake/alert/vital/active and a rating of 7 indicates the greatest feelings of sleepiness.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie A Cooper, PhD, Principal Investigator — University of Georgia
Locations (1):
- University of Georgia- Department of Foods and Nutrition, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
The plan is to share group averages through publication.

REFERENCES:
- [Derived] Guadagni AJ, Prater MC, Paton CM, Cooper JA. Cognitive function in response to a pecan-enriched meal: a randomized, double-blind, cross-over study in healthy adults. Nutr Neurosci. 2025 Sep;28(9):1075-1092. doi: 10.1080/1028415X.2025.2461018. Epub 2025 Feb 13. PMID 39945748
- [Derived] Prater MC, Guadagni AJ, Cooper JA. Postprandial appetite responses to a pecan enriched meal: A randomized crossover trial. Appetite. 2024 Oct 1;201:107598. doi: 10.1016/j.appet.2024.107598. Epub 2024 Jul 4. PMID 38971424